CLINICAL TRIAL: NCT07229196
Title: Clinical Trial in Hypertensive Patients Comparing Two Cardiorespiratory Exercise Protocols, Low-volume Sprint Interval Training (SIT) Versus Moderate-intensity Continuous Training (MICT), to Evaluate Decreases in Ambulatory Blood Pressure and Other Clinical Variables.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unidad Enfermedades Cardiometabolicas- Hospital Interzonal General Agudos San Martin de La Plata (Other)
Responsible Party: Principal Investigator, Julian Minetto, Physican, Unidad Enfermedades Cardiometabolicas- Hospital Interzonal General Agudos San Martin de La Plata
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSMLP2025/178
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Hypertension (HTN)
Keywords: hypertension; exercise; low-volume sprint interval training; moderate-intensity continuous training; High-Intensity Interval Training
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, parallel-group clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MICT group: Continuous cycling at 50-70% of VO₂max, 15-30 minutes per session (Active Comparator): MICT group: Continuous cycling at 50-70% of VO₂max, 15-30 minutes per session
  Interventions: Behavioral: MICT group: Continuous cycling at 50-70% of VO₂max, 15-30 minutes per session.
- SIT group: 2-4 maximal 20-30-second cycling sprints (≥100% VO₂max) with recovery intervals (2-4 min) (Experimental): SIT group: 2-4 maximal 20-30-second cycling sprints (≥100% VO₂max) with recovery intervals (2-4 min), total duration ≤15 minutes per session.
  Interventions: Behavioral: SIT group: 2-4 maximal 20-30-second cycling sprints (≥100% VO₂max) with recovery intervals (2-4 min), total duration ≤15 minutes per session.

INTERVENTIONS:
Behavioral: SIT group: 2-4 maximal 20-30-second cycling sprints (≥100% VO₂max) with recovery intervals (2-4 min), total duration ≤15 minutes per session. — SIT group: 2-4 maximal 20-30-second cycling sprints (≥100% VO₂max) with recovery intervals (2-4 min), total duration ≤15 minutes per session.
  Three times per week for 12 weeks
  Arms: SIT group: 2-4 maximal 20-30-second cycling sprints (≥100% VO₂max) with recovery intervals (2-4 min)
Behavioral: MICT group: Continuous cycling at 50-70% of VO₂max, 15-30 minutes per session. — MICT group: Continuous cycling at 50-70% of VO₂max, 15-30 minutes per session. three times per week for 12 week
  Arms: MICT group: Continuous cycling at 50-70% of VO₂max, 15-30 minutes per session

SUMMARY:
This randomized clinical trial aims to compare two cardiorespiratory exercise training protocols - Sprint Interval Training (SIT), characterized by short, maximal-intensity efforts, versus Moderate-Intensity Continuous Training (MICT) - in patients with arterial hypertension. The primary objective is to evaluate the impact of both interventions on 24-hour ambulatory systolic blood pressure (ABPM) after a 12-week training period.

Secondary outcomes include diastolic, daytime, and nighttime blood pressure, metabolic and hemodynamic parameters, body composition, and serum myokine levels (IL-6 and α-CGRP).

Participants aged 30-59 years with diagnosed hypertension but without high cardiovascular risk will be recruited from the Cardio-Metabolic Disease Unit of Hospital San Martín (La Plata, Argentina). After a two-week familiarization period, eligible participants will be randomized to SIT or MICT groups.

The intervention will last 12 weeks, with three supervised sessions per week. The study will provide valuable information about the effectiveness, safety, and clinical applicability of brief, high-intensity exercise for blood pressure control in hypertensive patients.

DETAILED DESCRIPTION:
Introduction

Cardiovascular disease remains the leading cause of mortality worldwide, with hypertension as a major modifiable risk factor. Exercise is a key non-pharmacological strategy for blood pressure management. While moderate-intensity continuous training (MICT) is well established, Sprint Interval Training (SIT) - characterized by short (10-30 s) bursts of maximal effort - has shown promising metabolic and cardiovascular benefits with significantly shorter session durations.

Despite growing interest, few clinical trials have evaluated SIT in hypertensive populations using ambulatory blood pressure monitoring (ABPM), which provides better prognostic information than office measurements. Furthermore, the biological mechanisms underlying exercise-induced benefits may involve myokines such as interleukin-6 (IL-6) and α-calcitonin gene-related peptide (α-CGRP), both associated with improved cardiometabolic health.

Objectives

Primary objective:

To compare the effect of SIT versus MICT on 24-hour systolic ambulatory blood pressure after 12 weeks of structured exercise.

Secondary objectives:

Assess changes in diastolic, daytime, and nighttime ambulatory blood pressure.

Evaluate office BP, anthropometric variables (weight, waist circumference, body fat percentage), and metabolic profile (lipids, glucose, TG/HDL ratio).

Assess changes in maximal oxygen consumption (VO₂max), non-invasive hemodynamic parameters, and handgrip strength.

Determine post-training serum concentrations of IL-6 and α-CGRP as biomarkers of exercise response.

Analyze acute hemodynamic responses and adherence to training.

Materials and Methods

Design:

Open-label, randomized, parallel-group clinical trial with pre- and post-intervention evaluations.

Population:

Hypertensive adults (30-59 years) attending the Cardio-Metabolic Disease Unit of Hospital San Martín (La Plata, Argentina).

Inclusion criteria:

Confirmed hypertension (treated or untreated).

BMI 18.5-34.9 kg/m².

Exclusion criteria:

Office BP ≥160/100 mmHg.

Diabetes, chronic kidney disease (eGFR <60 mL/min), coronary or cerebrovascular disease, pregnancy, or severe comorbidities.

Intervention:

Participants undergo a 2-week familiarization phase before randomization into two groups:

MICT group: Continuous cycling at 50-70% of VO₂max, 15-30 minutes per session.

SIT group: 2-4 maximal 20-30-second cycling sprints (≥100% VO₂max) with recovery intervals (2-4 min), total duration ≤15 minutes per session.

Both groups train three times per week for 12 weeks, under professional supervision. Blood pressure, heart rate, and oxygen saturation will be monitored during sessions for safety.

Evaluations:

At baseline and post-intervention:

Office and 24-hour ABPM measurements.

Anthropometry and laboratory tests (lipid profile, glucose, IL-6, α-CGRP via ELISA).

Impedance cardiography and pulse wave velocity for non-invasive hemodynamics.

Graded exercise test to determine VO₂max.

Handgrip strength test.

Sample size:

A total of 14-20 participants (7-10 per group) are required to detect a 5 mmHg difference in 24-hour systolic BP with 80% power and α=0.05.

Statistical analysis:

Between-group comparisons will use t-tests or Wilcoxon rank-sum tests depending on data distribution. Within-group pre/post differences will be analyzed with paired tests. Analyses will follow the intention-to-treat principle, with additional per-protocol analysis for participants achieving ≥75% adherence.

Ethics:

The study is classified as minimal risk and adheres to the Declaration of Helsinki (2024). Approved by the Ethics Committee of Hospital San Martín de La Plata (Reg. No. 070/2019). All participants will provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes between 30-59 years of age who meet the definition of hypertension.

Hypertension will be defined as:

1. Those patients who report a history of hypertension and are under pharmacological treatment for it (Angiotensin Converting Enzyme Inhibitors/Angiotensin II Receptor Antagonists/Calcium Channel Blockers/Thiazide Diuretics/Beta Blockers) at the time of the evaluation.

   OR
2. Patients who report a history of hypertension during the evaluation and who, without pharmacological treatment, have average levels ≥140/90 mmHg will also be considered hypertensive.

Exclusion Criteria:

* Extreme body mass index (BMI) <18.5 and ≥35.
* Patients with office blood pressure readings ≥160/100 mmHg.
* Patients with high cardiovascular risk conditions such as type II diabetes, chronic kidney disease (<60 milliseconds), history of cerebrovascular disease, coronary artery disease, peripheral arterial disease, or heart failure (Framingham Criteria clinical diagnosis).
* Pregnant or postpartum women up to 3 months old.
* Patients with psychophysical limitations that make exercise difficult.
* Patients with a history of active malignant neoplastic disease under treatment.

Elimination Criteria

-Patients whose pharmacological treatment is initiated or modified during the follow-up after 3 months.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the differences between both exercise protocols in 24-hour systolic ambulatory blood pressure (ABPM) values after the 12-week programmed exercise | after the 12-week programmed exercise

SECONDARY OUTCOMES:
To evaluate the differences between both exercise protocols in 24-hour diastolic ambulatory blood pressure (ABPM) values after the 12-week programmed exercise | after the 12-week programmed exercise
To evaluate the differences between both exercise protocols in daytime and nighttime ambulatory ABPM values after the 12-week programmed exercise. | after the 12-week programmed exercise
To evaluate the differences in other clinical characteristics such as office SBP and DBP, weight, waist circumference, and percentage of body fat through skinfold thickness measurements after the 12-week programmed exercise. | after the 12-week programmed exercise.
To evaluate the differences between both exercise protocols in insulin resistance and lipid profile parameters (TG/HDL, TG/glycemia, glycemia, LDL) after the 12-week programmed exercise | after the 12-week programmed exercise
To evaluate the differences between both exercise protocols in maximal oxygen uptake capacity (Vo2max) after the 12-week programmed exercise | after the 12-week programmed exercise
To evaluate the differences between both exercise protocols in noninvasive hemodynamics (peripheral resistance/cardiac index) after the 12-week programmed exercise | after the 12-week programmed exercise
To determine plasma levels of interleukin-6 and calcitonin gene-related peptide alpha after the 12-week programmed exercise. | after the 12-week programmed exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Espeche, Principal Investigator — Hospital Interzonal General San Martin; Julian Minetto, Physican, Principal Investigator — Hospital interzonal general agudos San Martin de La Plata; Matias Santamaria, Principal Investigator — Hospital interzonal general agudos San Martin de La Plata
Locations (1):
- Hospital Interzonal General San Martin La Plata, La Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
Potentially yes, given the conditions of anonymity as well as the instances of prior agreement and grounds for the reques